CLINICAL TRIAL: NCT05534958
Title: Assessing the Diagnostic Accuracy of a Three One-minute Tests of Verbal Fluency, Using Artificial Intelligence, in Detecting Mild Cognitive Impairment and Early Dementia.
Brief Title: UK Validation of the Automated "AcceXible" Speech Analysis Software
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Accexible (Industry)
Collaborators: Cornwall Partnership NHS Foundation Trust (Network)
Responsible Party: Sponsor
Other Study IDs: AcceXible-Healthy,MCI,Dementia
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-08

CONDITIONS: Mild Cognitive Impairment and Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy
  Interventions: Device: Accexible
- Mild Cognitive Impairment
  Interventions: Device: Accexible
- Early Dementia
  Interventions: Device: Accexible

INTERVENTIONS:
Device: Accexible — Speech Analysis

SUMMARY:
Dementia, especially dementia caused by Alzheimer's disease, is considered one of the most severe health problems of our time. It is currently known that the disease begins many years before clinical symptoms appear. The sooner the patient is diagnosed, the sooner the patient will be in a position to prevent further deterioration.

A recent orientation is the analysis of language in relation to the description of images with a high and varied semantic and emotional content. It can be studied that changes in the description of an image check if these changes are associated with the evolution of a person with probable impairment both in memory and cognitive as well as emotional, psychiatric, behavioral and even in their interaction with environmental factors especially those associated with socialization and loneliness.

The present study has the objective of validating a digital method for detection and follow-up of patients with mild cognitive impairment (MCI) or dementia in a memory clinic setting.

ELIGIBILITY:
Inclusion Criteria for patients:

* Adult patients 55+ years of age with suspected MCI or diagnosis of dementia referred into secondary care memory clinic by their General Practitioner.
* Have English as first language (able to speak and understand verbal messages).
* Patients must have agreed to participate in the study and have voluntarily signed the informed consent.

Inclusion Criteria for healthy volunteers:

* Healthy older adults (55+ years of age), without a diagnosis neurological, or psychiatric disorders or any clinical evidence of cognitive decline.
* Have English as first language (able to speak and understand verbal messages).
* Controls must have agreed to participate in the study and have voluntarily signed the informed consent.

Exclusion Criteria for patients:

* To have received a diagnosis of a significant psychiatric disorder or other cognitive impairment not due to neurodegeneration.
* To have significant vision problems that would affect the ability to perceive visual stimuli.
* To have significant hearing problems that would affect the ability to understand verbal cues.
* To be unable to give informed consent to participate in the study.

Exclusion Criteria for healthy volunteers:

* Objective evidence of significant cognitive decline in any one domain.
* Score of <88 on ACE-III cognitive testing.

Ages: 55 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Sample:
  Cases: 125 adult patients >55 years with suspected MCI or diagnosis of dementia referred to memory clinic.
  Controls: 125 healthy adult patients >55 years without a diagnosis of MCI and without subjective cognitive complaints.
Sampling Method: Probability Sample
Enrollment: 248 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of Accexible's digital screening battery | An average of 1 year
  Measure the odds that a patient has MCI or dementia measured by vocal biomarkers

SECONDARY OUTCOMES:
Correlation of Accexible's test battery with the ACE III | An average of 1 year
  Comparison of Accexible's test battery with ACE III diagnostic predictive value at various cut-off points (e.g. 82 and 88 for ACE III)

CONTACTS AND LOCATIONS:
Locations (1):
- Cornwall Partnership NHS Foundation Trust, Cornwell, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided